CLINICAL TRIAL: NCT00663039
Title: Effects of Oxytocin Nasal Spray on Social Affiliation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, MPRC, L. Elliot Hong, M.D., University of Maryland, Baltimore
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: HP-00043595; P50MH082999 (NIH)
Record Dates: First submitted 2008-04-17; First posted 2008-04-21 (Estimated); Results first posted 2018-12-13 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Eye movements; phenotype; biochemical; relatives
MeSH Terms: conditions — Schizophrenia | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin, then Placebo (Experimental): Participants first received 24IU of Oxytocin administered intranasally with 6 total sprays (three in each nostril) on the morning and at midday of one study visit. Then, after at least month the participants returned for a second study day and received placebo.
  Interventions: Drug: Oxytocin
- Placebo, then Oxytocin (Experimental): Participants first received a placebo (saline nasal spray) administered intranasally with 6 total sprays (three in each nostril) on the morning and at midday of one study visit. Then, after at least month the participants returned for a second study day and received Oxytocin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — 24 IU oxytocin (or Placebo) in a total of 6 puffs (3 puffs per nostril)
  Other Names: Pitocin; Syntocinon
  Arms: Oxytocin, then Placebo
Drug: Placebo — Single dose (plus a booster dose) drug probe study using intranasal placebo
  Arms: Placebo, then Oxytocin

SUMMARY:
Schizophrenia is a complex and heritable disorder that encompasses several clinical symptom domains and functional impairments. Existing treatments of schizophrenia, although effective against positive symptoms, fail to benefit negative symptoms, the focus of the current protocol. One of the strategies of novel drug development depends on identifying heritable physiological deficits that mark the disease liability and are thought to occur along the causal pathway of negative symptoms. These heritable physiological deficits are often found in the biological relatives of schizophrenia proband; particularly those who have schizophrenia related personality styles [defined by schizophrenia spectrum personalities (SSP) in the diagnostic system], even though they do not have the full-blown illness. The current protocol will pilot a strategy of targeting biomarkers of negative symptoms using intranasal oxytocin in relatives of schizophrenia patients. The drug probe studies in such non-clinical sample have several advantages including the absence of other drug treatment that may modulate the response, and the lack of generalized deficits causing problems with task comprehension/engagement that may mute the therapeutic signal. In addition, finding of efficacy of the experimental drug on the target physiological deficit and the associated symptoms has clinical implications on its own rights. This is because about 25% of subjects with schizophrenia spectrum personality disorders experience serious functional impairments.

Oxytocin is an extensively used drug, which is well tolerated with few serious side effects. Several lines of evidence suggest its putative role in the treatment of negatives symptoms, particularly a lack of social drive and related symptoms.

DETAILED DESCRIPTION:
The current study will examine the effects of intranasal oxytocin on physiological/cognitive markers of negative symptoms in 24 participants with schizophrenia spectrum traits. Subjects will be tested in two one-day studies carried out at least a month apart. Subjects will receive a 24 IU dose of intranasal oxytocin (or placebo) followed by a battery of cognitive/neurophysiological tests administered 50 minutes later completed over the next 155 minutes. A second dose of the drug (oxytocin or placebo) will be administered 2 hours after the 1st in order to maintain therapeutic plasma levels and to complete all testing.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female subjects between ages of 18-64 years
* The presence of 3 or more SSP symptoms (at least 2 of the SSP symptoms will be negative symptoms as defined by the schizoid traits)
* The presence of visuo-spatial working memory impairment as defined by error in the oculomotor delayed response (ODR) task of more than 0.5 SD above the mean values in healthy control subjects
* Relative of an individual with schizophrenia, schizo-affective, or schizophreniform disorder
* Able to provide written informed consent. Females are excluded due to risk of discomfort and unblinding due to potential uterine cramps induced by oxytocin.

Exclusion Criteria:

* Subjects meeting criteria for a life-time diagnosis of any one of the DSM IV, Axis I psychotic disorders (exceptions being a single past episode of major depressive disorder with psychotic features or psychotic symptoms associated with substance abuse with the substance abuse ending 6-months prior to study participation) (this is for the SSP recruitment)
* Subjects meeting DSM-IV criteria for current alcohol or substance dependence (other than nicotine) within the last 6 months or DSM-IV criteria for alcohol or substance abuse (other than nicotine) within the last month
* Medical conditions that preclude participation in drug trials or assessments of outcome measures (including significant brain, cardiac, liver, lung, endocrinological or metabolic disorders)
* Received any investigational drug in the preceding four weeks.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2009-10 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L E Hong, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Maryland Psychiatric Research Center, Catonsville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxytocin, Then Placebo | Placebo, Then Oxytocin
Started | 14 | 13
Completed | 10 | 9
Not Completed | 4 | 4

BASELINE CHARACTERISTICS:
Population: Total participants that completed screening and considered eligible for study participation.
Groups:
- All Study Participants: Participants who were screened and met inclusion/exclusion criteria for the study.
Arm/Group | All Study Participants
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 8
  More than one race | 1
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Social Affiliation Measured by Social Affiliative Role Play
Description: In a videotaped session, research staff engages the participant in social interaction based on a role play. The tape is rated on social skills and on Positive and Negative Affect Scale. Participants are rated on a 5 point Likert scale ranging from very poor (1) to Very Good (5).
Time Frame: 30 minutes
Population: Of the 27 ppts that were screened and deemed eligible for study participation, only 19 completed testing while receiving oxytocin and only 18 complete testing while receiving placebo.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Oxytocin: Oxytocin Oxytocin: 24 IU oxytocin in a total of 6 puffs (3 puffs per nostril) administer at two intervals during 1 study visit.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 19 | 18
units on a scale
  Overall Affect | 4.026 (0.656) | 4.111 (0.583)
  Overall Social Skill | 4.079 (0.854) | 4.194 (0.622)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Comparison of Overall Affect Scores between Oxytocin and Placebo Arms; Test type: Superiority; p = 0.758, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Oxytocin vs Placebo; Comparison of Overall Social Skill scores between Oxytocin and Placebo arms; Test type: Superiority; p = 0.779, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Hopkins Verbal Learning Test (HVLT)
Description: HVLT comes in 6 different forms. Forms 4 and 5 were used for this study with one form administered on the first study day and the other on the second and were counterbalanced between subjects. Each form contains 12 nouns, four words each from one of three semantic categories, to be learned over the course of three learning trials.
Time Frame: 15 minutes
Population: Analyzable data for secondary outcomes was not available for some participants.
Measure: Mean (Standard Deviation); unit: Number of correct responses
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 16 | 14
Number of correct responses
  Hopkins Verbal Learning Test Trial1 | 6.19 (2.23) | 6.57 (1.79)
  Hopkins Verbal Learning Test Trial2 | 8.56 (1.93) | 9.36 (1.78)
  Hopkins Verbal Learning Test Trial3 | 10.12 (2.03) | 10.57 (1.40)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Comparison of HVLT Trial 1 scores between Oxytocin and Placebo Arms; Test type: Superiority; p = 0.578, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Oxytocin vs Placebo; Comparison of HVLT Trial 2 scores between Oxytocin and Placebo Arms; Test type: Superiority; p = 0.28, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Oxytocin vs Placebo; Comparison of HVLT Trial 3 scores between Oxytocin and Placebo Arms; Test type: Superiority; p = 0.707, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Trust Game
Description: Participants competed in a social trust game in which they are paired with a partner (the computer program). Over the course of 24 rounds the participant can offer up to $10 to their partner. The partner can either accept the offer, in which case the total amount offered is split equally between the participant and their partner (i.e. $10 is split into $5 each). Or the partner can reject the offer and receive an portion of the total offer for themselves and give the participant nothing ($0). The total amount of money that can be offered ranges from $0-240.
Time Frame: 20 minutes
Population: Analyzable data for secondary outcomes was not available for some participants.
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 16 | 14
Dollars | 112.5 (60) | 134.5 (68.5)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Comparison of the total amount of money offered during the trust game between the Oxytocin and Placebo arms; Test type: Superiority; p = 0.391, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: RVIP Reaction Times
Description: Rapid Visual Information Processing (RVIP) measures primarily sustained attention but perhaps also working memory. The task was continuous stimuli presentation of a stream of single digits (from 1 to 9) presented in the center of the computer monitor at a rate of 1/600milliseconds; the subjects respond when they see a target sequence of 3 odds or 3 even digits in a consecutive sequence. Two target sequences are separated by a minimum of 5 and maximum of 30 non-target digits
Time Frame: 25 minutes
Population: Analyzable data for secondary outcomes was not available for some participants.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 16 | 14
milliseconds
  RVIP Practice Mean Target Reaction Time | 563 (103) | 586 (110)
  RVIP First Half Mean Target Reaction Time | 588 (104.7) | 574.4 (82.9)
  RVIP Practice Mean False Alarms Reaction Time | 306.9 (49.5) | 277.1 (104.4)
  RVIP First Half Mean False Alarms Reaction Time | 302 (115) | 228 (138)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Comparison of RVIP Practice Mean Target Reaction Time between Oxytocin and Placebo arms; Test type: Superiority; p = 0.559, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Oxytocin vs Placebo; Comparison of RVIP First Half Mean Target Reaction Time between Oxytocin and Placebo arms; Test type: Superiority; p = 0.858, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Oxytocin vs Placebo; Comparison of RVIP Practice Mean False Alarms Reaction Time between Oxytocin and Placebo arms; Test type: Superiority; p = 0.514, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Oxytocin vs Placebo; Comparison of RVIP First Half Mean False Alarms Reaction Time between Oxytocin and Placebo arms; Test type: Superiority; p = 0.088, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Rapid Visual Information Processing Test (RVIP)
Description: RVIP measures primarily sustained attention but perhaps also working memory. The task was continuous stimuli presentation of a stream of single digits (from 1 to 9) presented in the center of the computer monitor at a rate of 1/600ms; the subjects respond when they see a target sequence of 3 odds or 3 even digits in a consecutive sequence. Two target sequences are separated by a minimum of 5 and maximum of 30 non-target digits. There are a total of 48 target sequences during each test block. The number of correctly Identified target sequences or hits is recorded, as well as, false alarms (incorrectly identified target sequences) and reaction times.
Time Frame: 25 minutes
Population: Analyzable data for secondary outcomes was not available for some participants.
Measure: Mean (Standard Deviation); unit: Number of responses
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 16 | 14
Number of responses
  RVIP Practice Mean Target Hits | 16.40 (8.58) | 19.15 (7.45)
  RVIP First Half Mean Target Hits | 17.80 (6.52) | 21.62 (6.99)
  RVIP Practice Mean False Alarms | 15.9 (16.5) | 10.2 (12.0)
  RVIP First Half Mean False Alarms | 14.7 (19.4) | 12.2 (15.5)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Comparison of RVIP Practice Mean Target Hits between Oxytocin and Placebo arms; Test type: Superiority; p = 0.296, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Oxytocin vs Placebo; Comparison of RVIP First Half Mean Target Hits between Oxytocin and Placebo arms; Test type: Superiority; p = 0.136, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Oxytocin vs Placebo; Comparison of RVIP Practice Mean False Alarms between Oxytocin and Placebo arms; Test type: Superiority; p = 0.47, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Oxytocin vs Placebo; Comparison of RVIP First Half Mean Target Hits between Oxytocin and Placebo arms; Test type: Superiority; p = 0.702, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Brief Assessments of Cognition for Schizophrenia
Description: The BACS Symbol Coding subtest will be used to assess processing speed, and the demographically corrected T score, will be used for data analysis. This test requires less than 5 minutes to administer and provides a highly reliable measure of processing speed. There are nine symbols code 1 through 9. Participants are given 90 seconds to match a series of these symbols with their corresponding number. The total correct matches is the participants score. Scores range from 0-110.
Time Frame: 5 minutes
Population: Analyzable data for secondary outcomes was not available for some participants.
Measure: Mean (Standard Deviation); unit: Number of correct responses
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 16 | 14
Number of correct responses | 45.6 (13.8) | 47.7 (14.3)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Comparison of Brief Assessments of Cognition for Schizophrenia scores between the Oxytocin and Placebo arms; Test type: Superiority; p = 0.451, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Brief Smell Identification Test
Description: The Brief Smell Identification Test (B-SIT) is a 5-minute, 12-item screening test. Participants try to identify 12 different odors with four multiple choice options given for each odor.
Time Frame: 5 minutes
Population: Analyzable data for secondary outcomes was not available for some participants.
Measure: Mean (Standard Deviation); unit: Number of correct responses
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 16 | 14
Number of correct responses | 10.06 (1.53) | 10.14 (1.10)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Superiority; p = 0.9, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Reading the Mind in the Eyes
Description: A 30 item task presents a picture of a person's eyes and the participant is ask to determine the person's mental state from 4 multiple choice options.
Time Frame: 10 minutes
Population: Analyzable data for secondary outcomes was not available for some participants.
Measure: Mean (Standard Deviation); unit: Number of correct responses
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 16 | 14
Number of correct responses | 24.40 (6.06) | 24.54 (5.78)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Comparison of Reading the Mind in the Eyes total scores between Oxytocin and Placebo arms; Test type: Superiority; p = 0.946, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Facial Affect Recognition
Description: This computer administered test includes 40 color photographs of four universal emotions (happy, sad, angry, and fearful) balanced for the posers gender, age, and ethnicity, including four low intensity and four high-intensity facial expressions of each emotion, plus 8 neutral faces. The stimuli are presented in random order and subjects are asked to identify which stimuli were presented to them at the end. Performance on this test correlates with negative symptom severity.
Time Frame: 10 minutes
Population: Analyzable data for secondary outcomes was not available for some participants.
Measure: Mean (Standard Deviation); unit: Number of responses
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 16 | 14
Number of responses
  Facial Affect Recognition Total | 29.79 (4.69) | 34.08 (5.33)
  Facial Affect Recognition Hits | 12.86 (5.36) | 15.46 (4.22)
  Facial Affect Recognition False Alarms | 6.71 (4.51) | 5.38 (3.01)
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Comparison the Facial Affect Recognition Total scores between Oxytocin and Placebo arms; Test type: Superiority; p = 0.016, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Oxytocin vs Placebo; Comparison the Facial Affect Recognition Hits between Oxytocin and Placebo arms; Test type: Superiority; p = 0.185, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Oxytocin vs Placebo; Comparison the Facial Affect Recognition False Alarms between Oxytocin and Placebo arms; Test type: Superiority; p = 0.404, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Collected over the course of 2 approximately 8 hour study days.
Description: The Side Effect Checklist was used
Groups:
- Oxytocin: Oxytocin administered on study
- Placebo: Placebo administered on study day
Arm/Group | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 3/19 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin (N=19) | Placebo (N=18)
Dizziness (General disorders) | 1 (1) | 0 (0) — Participant became slightly dizzy during testing.
Drowsiness (General disorders) | 1 (1) | 0 (0) — Participant reported feeling drowsy during testing
Euphoria (General disorders) | 1 (1) | 0 (0) — Participant reported a brief state of euphoria following study drug administration

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No